CLINICAL TRIAL: NCT01442987
Title: Efficacy and Safety of Coadministered Irbesartan and Atorvastatin in Patients With Hypertension and Hyperlipidemia
Brief Title: Efficacy and Safety of Irbesartan and Atorvastatin in Hypertension and Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HM-IBAT-301
Record Dates: First submitted 2011-07-01; First posted 2011-09-29 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Hypertension; Hyperlipidemia
Keywords: Irbesartan; Atorvastatin; Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Irbesartan/Atorvastatin A (Experimental)
  Interventions: Drug: Irbesartan/Atorvastatin A
- Irbesartan (Active Comparator)
  Interventions: Drug: Irbesartan
- Atorvastatin A (Active Comparator)
  Interventions: Drug: Atorvastatin A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Irbesartan/Atorvastatin B (Experimental)
  Interventions: Drug: Irbesartan/Atorvastatin B
- Atorvastatin B (Active Comparator)
  Interventions: Drug: Atorvastatin B

INTERVENTIONS:
Drug: Irbesartan/Atorvastatin A — once daily, P.O. 8week
  Other Names: HCP0912 A
  Arms: Irbesartan/Atorvastatin A
Drug: Irbesartan — once daily, P.O. 8week
  Arms: Irbesartan
Drug: Atorvastatin A — once daily, P.O. 8week
  Arms: Atorvastatin A
Drug: Placebo — once daily, P.O. 8week
  Arms: Placebo
Drug: Irbesartan/Atorvastatin B — once daily, P.O. 8week
  Other Names: HCP0912 B
  Arms: Irbesartan/Atorvastatin B
Drug: Atorvastatin B — once daily, P.O. 8week
  Arms: Atorvastatin B

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of coadministered Irbesartan and Atorvastatin in patients with hypertension and hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 75 years
* Signed informed consent

Exclusion Criteria:

* At screening, SPB ≥ 180mmHg or DBP ≥ 110mmHg or LDL-C > 250mg/dL or TG ≥ 400mg/dL
* Has a history of hypersensitivity to Angiotensin Ⅱ receptor blocker or HMG-CoA reductase inhibitor or component of this drug
* Has a history of multi-drug allergy

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to 8 week in LDL-Cholesterol | baseline and 8 week
Change from baseline to 8 week in Blood Pressure. | baseline and 8 week

SECONDARY OUTCOMES:
Percentage of patients reaching treatment goals according to NCEP ATP III Guideline and Blood pressure responder rate according to JNC VII Guideline. | week 8

CONTACTS AND LOCATIONS:
Overall Officials: Byeong Hee Oh, M.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- 16 institutions including Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim SH, Jo SH, Lee SC, Lee SY, Yoon MH, Lee HL, Lee NH, Ha JW, Lee NH, Kim DW, Han GR, Hyon MS, Cho DG, Park CG, Kim YD, Ryu GH, Kim CH, Kim KS, Chung MH, Chae SC, Seung KB, Oh BH. Blood Pressure and Cholesterol-lowering Efficacy of a Fixed-dose Combination With Irbesartan and Atorvastatin in Patients With Hypertension and Hypercholesterolemia: A Randomized, Double-blind, Factorial, Multicenter Phase III Study. Clin Ther. 2016 Oct;38(10):2171-2184. doi: 10.1016/j.clinthera.2016.09.005. Epub 2016 Oct 12. PMID 27742464